CLINICAL TRIAL: NCT01846845
Title: Prosthetic Socket System: Pilot Assessment
Brief Title: Evaluation of a Novel Transfemoral Prosthetic Socket System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ohio Willow Wood (Industry)
Collaborators: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: VA-2012-Aim3; VA118-12-C-0038 (Other Grant/Funding Number: Veterans Affairs Innovation Initiative)
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2013-06

CONDITIONS: Lower Limb Amputation
Keywords: Amputee

ARMS (2):
- Conventional TF Socket System (Active Comparator): Conventional Prosthetic Transfemoral Socket System
  Interventions: Device: Conventional Prosthetic Transfemoral Socket System
- Novel TF Socket System (Experimental): Novel Prosthetic Transfemoral Socket System
  Interventions: Device: Novel Prosthetic transfemoral socket system

INTERVENTIONS:
Device: Conventional Prosthetic Transfemoral Socket System — Conventional transfemoral may include an ischial containment socket, a pin suspension socket, and/or suction suspension socket
  Other Names: Ischial Containment; Pin Transfemoral Socket; Suction Transfemoroal Socket; Above the knee (AK) socket
  Arms: Conventional TF Socket System
Device: Novel Prosthetic transfemoral socket system — Prosthetic socket that incorporates lower socket trim-lines and transfemoral vacuum suspension
  Arms: Novel TF Socket System

SUMMARY:
The purpose of the study is to evaluate residual limb circulation and skin health associated with the use of a novel prosthetic transfemoral socket system. A conventional prosthesis will be compared to the novel transfemoral socket system.

DETAILED DESCRIPTION:
Conventional transfemoral socket designs impose an array of limitations on transfemoral amputee patients. Flexion, extension, and abduction are considerably impaired and end basic functions like sitting are usually uncomfortable or even painful. An alternative socket design that lowers the socket trim-lines and still provides structural support would greatly improve the socket comfort for transfemoral amputees.

ELIGIBILITY:
Inclusion Criteria:

* Consenting Adult
* Unilateral transfemoral amputee
* Currently suing a liner with prosthesis
* Uses a prosthesis to ambulate
* Ability to read, write, and understand English
* Available during regular business hours for appointments

Exclusion Criteria:

* Impaired contra lateral leg
* Ambulates with the aid of an additional assistive device (e.g. walker, cane, etc.)
* Diagnosis of renal failure
* Smoker

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Laser Doppler flowmetry tissue perfusion values | 1 month
  Change from baseline in Laser Doppler flowmetry tissue perfusion values at 1 month

SECONDARY OUTCOMES:
Laser speckle flowmetry tissue perfusion values | 1 month
  Change from baseline in laser speckle flowmetry tissue perfusion values at 1 month
Hyperspectral Imaging Tissue Oxygen Saturation (StO2%) | 1 month
  Change from baseline in hyperspectral imaging StO2% at 1 month
Trans-Epidermal Water Loss values | 1 month
  Change from baseline in trans-epidermal water loss values at 1 month
Surface electrical capacitance values | 1 month
  Change from baseline in surface electrical capacitance values at 1 month
Elasticity (cutometry) values | 1 month
  Change from baseline in elasticity values at 1 month
Torsional Ballistometry values | 1 month
  Change from baseline in torsional ballistometry values at 1 month

OTHER OUTCOMES:
Skin temperature values | 1 month
  Change from baseline in skin temperature values at 1 month
Prosthesis evaluation questionnaire (PEQ) | 1 month
  Change from baseline in prosthesis evaluation response at 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Gayle Gordillo, MD, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - The Ohio State University Davis Heart and Lung Research Institute, Columbus, Ohio
  - The Ohio Willow Wood Company, Mount Sterling, Ohio